CLINICAL TRIAL: NCT05913609
Title: IDE Clinical Study to Evaluate the Safety and Effectiveness of the Yaari Extractor for Management of Shoulder Dystocia
Brief Title: Safety and Effectiveness of the Yaari Extractor for Management of Shoulder Dystocia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FetalEase Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLT-005
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Dystocia
MeSH Terms: conditions — Shoulder Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Yaari Extractor group (Experimental): Prospective experimental arm
  Interventions: Device: Yaari Extractor
- Control group (No Intervention): Historical control arm - retrospective review of medical records at the same study sites

INTERVENTIONS:
Device: Yaari Extractor — The Yaari Extractor device is a single-use prescription device for neonatal extraction in deliveries that are complicated by shoulder dystocia. The Study Device consists of two curved, rigid plastic-coated metal Arms with Handles which are used for control of the device outside the body, and an elastic Engagement Element which conforms to the maternal and neonatal anatomy, and which is used for direct contact with the entrapped neonate within the birth canal.
  Arms: Yaari Extractor group

SUMMARY:
Prospective, multi-center, single arm with historical control, to verify the safety and effectiveness of the Yaari Extractor used by board certified or board eligible U.S. OB/GYN physicians in the management of shoulder dystocia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject 18 years of age or older at time of consent.
2. Subject planning on vaginal birth.
3. Singleton pregnancy in vertex presentation.
4. Full-term pregnancy having completed 37 weeks or more gestational weeks.
5. Able and willing to provide written informed consent prior to enrollment.
6. In the opinion of the Investigator, the subject has sufficient mental capacity to understand the informed consent form (ICF).
7. Subject with fetus experiencing shoulder dystocia as defined by ACOG Practice Bulletin 178 "Shoulder dystocia is most commonly diagnosed as failure to deliver the fetal shoulder(s) with gentle downward traction on the fetal head, requiring additional maneuvers to effect delivery."

Exclusion Criteria:

1. Patients who have undergone attempted delivery using ancillary standard of care maneuvers, to include first-line maneuvers (McRoberts ± suprapubic pressure with downward traction on the fetal head), prior to use of the Yaari Extractor. (NOTE: Hyperflexion of the hips or legs is allowed prior to and during use of the Yaari Extractor.)
2. Cesarean section is planned for the patient.
3. Obstetric contraindications to vaginal birth.
4. Subject carrying fetus with known significant chromosomal or structural anomalies.
5. Clinically estimated fetal weight ≥5kg in non-diabetic subjects.
6. Clinically estimated fetal weight ≥4.5kg in subjects with diabetes.
7. Subject has any general health condition or systemic disease that may represent, in the opinion of the Investigator, a potential increased risk associated with device use or pregnancy.
8. Bleeding disorders, such as thrombocytopenia, von Willebrand's disease, bleeding disorder currently using anticoagulation medication, etc.
9. Any maternal disease or disorder that precludes the subject from pushing effectively.
10. If the maternal cervix is not fully dilated.
11. If the fetal head is not completely out of the birth canal.
12. In the presence of a non-reducible nuchal cord.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of successful neonate deliveries with the Yaari Extractor device | immediately after the intervention
  First Primary Effectiveness Endpoint
Time interval (minutes) from the diagnosis of the shoulder dystocia until the neonate's delivery | immediately after the intervention
  Second Primary Effectiveness Endpoint
Maternal and neonatal adverse events | through study completion, an average of 5 days
  Primary Safety Endpoint

SECONDARY OUTCOMES:
Ease of Use 5 point Likert scale User Questionnaire | immediately after the intervention
  Secondary Effectiveness Endpoint

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Miami - Jackson Memorial, Miami, Florida
  - Rosemark WomenCare Specialist, Idaho Falls, Idaho
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No